CLINICAL TRIAL: NCT06743711
Title: Validation and Impact of Cardiorespiratory Fitness in Severe Mental Illness - the Heart in Mind Project
Status: Recruiting | Type: Observational
Sponsor: Bjorn H. Ebdrup (Other)
Collaborators: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other); VentriJect ApS (Industry)
Responsible Party: Sponsor-Investigator, Bjorn H. Ebdrup, Professor and consultant psychiatrist, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: H-24031121; 2023-0065 (Other Grant/Funding Number: Simon Fougner Hartmanns Familiefond); H-24031121 (Other: The Scientific Ethical Committees for the Capital Region of Denmark)
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Severe Mental Illness; Schizophrenia Spectrum & Other Psychotic Disorders; Bipolar Affective Disorder
Keywords: cardiorespiratory fitness; severe mental illness; cardiovascular disease; validation; physical activity; cardiopulmonary exercise test; non-exercise vo2max estimation; vo2max
MeSH Terms: conditions — Mental Disorders; Bipolar Disorder; Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Adults with severe mental illness in treatment with antipsychotic medications
- Healthy controls: Adults without present or previous mental illness, and no first-degree relatives with present or previous mental illness, matched to the patient group for gender, age, and BMI.

SUMMARY:
This project aims to evaluate feasibility, validity and clinically applicability to systematically measure fitness in patients with severe mental illness.

The research project is a validation study using a cross-sectional design. The project will include 50 people with severe mental illness and 25 healthy controls without present or previous mental illness. The protocol includes a baseline visit where three different ways of measure fitness will be carried out, and a 14-day period of physical activity monitoring.

DETAILED DESCRIPTION:
BACKGROUND Cardiorespiratory fitness (CRF) is a strong independent predictor of cardiovascular disease (CVD) and all-cause mortality in the general population. However, CRF is rarely considered or measured in psychiatric populations, despite people with severe mental illness (SMI) is a high-risk population of CVD and may suffer from premature death of up to 15-20 years.

AIM The aim of this project is to evaluate the feasibility, validity, and clinical relevance of CRF assessment in patients with SMI.

POPULATION 50 people with severe mental illness in treatment with antipsychotic medications and 25 healthy controls without present or previous mental illness matched for sex, age, and BMI will be included in the study.

METHODS This is a validation study with a cross-sectional design. The study includes a ~3 hour baseline visit and 14 days of physical activity monitoring.

Baseline Visit (D0) Physical health, body composition, vital signs, and non-exercise VO2max estimation by seismocardiography (SCG) will be carried out initially. Afterwards, psychopathology, substance use, and cognition will be assessed during an interview. Questionnaires regarding physical activity, fitness, quality of life, body image and self-esteem, and sleep will be completed by the participants.

Essential for the baseline visit, two fitness tests will be conducted. First, the revised Ekblom-Bak submaximal cycle-ergometer fitness test followed by a state-of-the-art graded cardiopulmonary exercise test to exhaustion. During both tests, oxygen uptake will be assessed with gas-exchange analysis equipment. After the baseline visit, participants will wear a physical activity sensor (SENS Motion(R)) for two weeks, and finish participation in the study with completion of questionnaires.

ELIGIBILITY:
Patients

Inclusion Criteria:

* 1) 18-45 years; 2) Diagnosis within schizophrenia spectrum or affective disorders (i.e. F2.x or F3.x according to ICD-10 classification); 3) current antipsychotic treatment for more than one month on a regular daily dose and 4) Able to give informed consent.

Exclusion Criteria:

* 1) Clinical or laboratory evidence of uncompensated medical disease; 2) Unstable psychiatric disorder; 3) Acute suicidal risk; 4) Planned hospitalization within the study period.

Healthy controls

Inclusion Criteria:

* 1) 18-45 years; 2) No psychiatric diagnosis or having first-degree relatives with psychiatric diagnoses; 3) able to give informed consent.

Exclusion Criteria:

* 1) Clinical or laboratory evidence of uncompensated medical disease; 2) Indication of psychiatric disorder.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited from inpatient and outpatient clinics in the Capital Region of Denmark. Furthermore, recruitment will also be carried out through two ongoing randomized controlled trials i) Value of gym-based exercise training for young adults with severe mental illness: A pragmatic, single-blinded, multicenter randomized controlled trial - the Vega trial (NCT05461885), and ii) Effectiveness of a pragmatic, metabolic care clinic for patients with severe mental illness (NCT06624462).
  Healthy controls will be recruited through announcements in the Capital Region of Denmark, through the webpages www.forsøgsperson.dk and www.forskningnu.dk and social media.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Validation of the revised Ekblom-Bak submaximal cycle-ergometer fitness test | At baseline visit (D0)
  The revised Ekblom-Bak submaximal cycle-ergometer fitness test (EBsub) will be carried out to estimate VO2max and validated against measured VO2max during a cardiopulmonary exercise test (CPET) including calculation of coefficient variation, limits of agreement, mean absolute percentage error, linear regression analyses for obtaining R-squared values and standard errors of the estimate, and Bland-Altman plotting.
  VO2max will be assessed during an incremental cycle protocol until exhaustion conforming to the state-of-the-art CPET. Oxygen consumption and carbon dioxide excretion rates will be measured using a "breath-by-breath" analysing system coupled to a fitted silicone mask, strapped around the participants head, covering nose and mouth (Vyntus CPX, Jaeger). VO2max will be defined as the average of the three highest oxygen consumption measurements.
  VO2max will be estimated with the EBsub conforming to the developing authors guidelines.

SECONDARY OUTCOMES:
Validation of non-exercise VO2max estimation by seismocardiography | At baseline visit (D0)
  Non-exercise VO2max estimation with seismocardiography (SCG) will be carried out to estimate VO2max and validated against measured VO2max during a cardiopulmonary exercise test (CPET) including calculation of coefficient variation, limits of agreement, mean absolute percentage error, linear regression analyses for obtaining R-squared values and standard errors of the estimate, and Bland-Altman plotting.
  VO2max will be assessed during an incremental cycle protocol until exhaustion conforming to the state-of-the-art CPET. Non-exercise VO2max estimation through SCG will be carried out with the Seismofit(R) (VentriJect, Denmark) device conforming to manifacturers instructions. Breifly, the Seismofit device will be mounted on the sternum, 2 cm proximal to the Xiphoid Process. Before estimation, age, height, weight, and sex of the participant is entered into the VentriJect app. The VO2max estimation lasts ~5min, including recording, data transfer, and signal processing.

OTHER OUTCOMES:
Physical activity | From baseline to study end after 14 days
  International Physical Activity Questionnaire (IPAQ) Physical Activity Vital Sign (PAVS) Accelorometry (SENS Motion(R))
Self-perceived fitness | At baseline visit and at study end after 14 days
  self-perceived cardiorespiratory fitness on a 5-point Likert scale rating (i.e., very poor, poor, fair, good, very good) to the question; How do you rate you own physical fitness?
Psychopathology | At baseline visit (D0)
  Psychopathology will be assessed with the Positive and Negative Syndrome Scale (PANSS), which provides a structured format for clinicians to evaluate symptom severity in people with psychotic symptoms and/or schizophrenia. Clinicians rate the severity of each symptom on a scale ranging from 1 (not present) to 7 (extremely severe).
Negative symptoms | At baseline visit (D0)
  Negative symptoms will be assessed with The Brief Negative Symptom Scale (BNSS), which is a standardized clinical assessment tool designed to measure the severity of negative symptoms in individuals with schizophrenia spectrum disorders. Developed as a concise complement to existing scales, the BNSS focuses specifically on assessing five domains of negative symptoms: blunted affect, alogia, anhedonia, asociality, and avolition. Each domain is evaluated through a series of items, with clinicians rating the severity of each symptom on a scale from 0 (absent) to 6 (severe).
Depressive symptoms | At baseline visit (D0)
  Depressive symptoms will be assessed with the modified Major Depression Index (mMDI), which is a refined assessment tool utilized in clinical and research settings to evaluate the severity of major depressive disorder (MDD) symptoms. This index, encompasses key domains of depressive symptomatology, including mood disturbances, cognitive impairments, vegetative symptoms, and psychomotor changes. The mMDI consists of a structured interview format of ten items on a scale of 1 (at no time) to 5 (most of the time).
Global cognition | At baseline visit (D0)
  Global cognition will be assessed with the Brief Cognitive Assessment Tool for Schizophrenia (B-CATS), which is a validated instrument taking approximately ten minutes employed in clinical and research contexts to evaluate cognitive functioning in individuals with schizophrenia spectrum disorders. Developed to efficiently assess cognitive domains relevant to schizophrenia, the B-CATS encompasses key areas such as attention, memory, executive function, and processing speed. The B-CATS includes four tests; 1) Digit Symbol Substitution, 2) Trail Making Test A, 3) Trail Making Test B, and 4) Animal Fluency, which together provides a measure of global cognitive functioning.
Sleep quality | At baseline visit (D0)
  Sleep quality will be assessed with the Brief Pittsburgh Sleep Quality Index (B-PSQI) is a shorter version of the PSQI, designed to provide a quick assessment of sleep quality and disturbances. It includes six items from the original PSQI, focusing on key aspects such as subjective sleep quality, sleep duration, and sleep disturbances.
Drug use | At baseline visit (D0)
  Drug use will be assessed with the Drug Use Disorders Identification Test (DUDIT), which is a validated screening tool designed to assess drug use and related problems in individuals aged 15-65. It consists of 11 items that cover various aspects of drug use, including frequency, quantity, and consequences of use on a 1 to 5 Likert scale. The total score provides an indication of the severity of drug-related problems, with higher scores indicating greater severity.
Alcohol use | At baseline visit (D0)
  Alcohol use will be assessed with The Alcohol Use Disorders Identification Test (AUDIT) is a widely used screening tool developed by the World Health Organization (WHO) to assess alcohol consumption patterns and identify individuals at risk of alcohol-related problems. The AUDIT covers three domains: alcohol consumption, alcohol dependence symptoms, and alcohol-related problems. The AUDIT consists of ten items, where each item scored on a Likert scale ranging from 0 to 4.
  The total score provides an indication of the severity of alcohol use and related issues, with higher scores indicating greater risk.
Smoking | At baseline visit (D0)
  Smoking will be assessed with the Fagerström Test for Nicotine Dependence (FTND), which is a validated assessment tool designed to measure the degree of nicotine dependence in tobacco users. The FTND comprises six items that assess various aspects of nicotine dependence, including the intensity of tobacco craving, the frequency of smoking, and the compulsion to smoke in specific situations. The total score provides a quantitative measure of nicotine dependence severity, with higher scores indicating greater dependence.
Quality of life | At baseline visit (D0)
  General quality of life, physical health, psychological, social relationships, environment will be assessed with the World Health Organization Quality of Life-Brief (WHOQOL-Bref) is a validated instrument developed by the World Health Organization (WHO) to assess individuals' quality of life across physical, psychological, social relationships, and environmental domains. Derived from the WHOQOL-100, the WHOQOL-Bref consists of 26 items that cover these four domains, providing an evaluation of subjective well-being. Respondents rate their perceptions of various aspects of life on a Likert scale, with higher scores indicating better quality of life.
Body weight, image, and self esteem | At baseline visit (D0)
  Body weight, image, and self esteem will be assessed with the Body Weight, Image, and Self-Esteem (B-WISE), which is a validated assessment tool designed to evaluate the interrelationship between body weight perception, body image dissatisfaction, and self-esteem. The B-WISE comprises 12 items, each item scored on a 1 to 3 Likert scale with higher scores indication poorer adjustment (i.e., never, sometimes, and all the time).
Anthropometrics | At baseline visit (D0)
  Anthropometrics including height and circumferences will be measured. Height will be assessed without shoes with a wall-mounted stadiometer and waist and hip circumference will be measured with measuring tape, both with a sensitivity of 0.1cm.
Body composition | At baseline visit (D0)
  Body composition will be assessed with a seca mBCA 514/515 bioelectrical impedance analysis (BIA) machine (SECA GmbH). Utilizing BIA technology, the Seca mBCA 514/515 measures the body's impedance to a small electrical current, which varies based on the amount of water and electrolytes present in different body compartments and tissue. By analyzing the impedance data and applying validated algorithms, the Seca MBCA estimates various components of body composition, including fat mass, fat-free mass, body water, and muscle mass. Additionally, it can estimate visceral adipose tissue when provided with waist circumference.
Blood pressure and resting heart rate | At baseline visit (D0)
  Blood pressure and resting heart rate will be assessed when the participant is resting and an average of three measurements with a digital blood pressure device (Rossmax) will be carried out.
Electrocardiogram | At baseline visit (D0)
  Electrocardiogram will be assessed with an electrocardiograph when the participant is resting and lying down.
Metabolic profile | At baseline visit (D0)
  Metabolic profile will be assessed by accessing the participant's medical record and using the latest blood sample analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn H Ebdrup, Professor and psychiatrist, Study Director — Mental Health Center Glostrup, Center for Neuropsychiatric Schizophrenia Research; Victor Sørensen, PhD student, Principal Investigator — Mental Health Center Glostrup, Centre for Applied Research in Mental Health Care & Center for Neuropsychiatric Schizophrenia Research
Locations (1):
- Mental Health Center Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Heart in Mind — https://www.psykiatri-regionh.dk/cnsr/current_projects/heartinmind/Sider/default.aspx